CLINICAL TRIAL: NCT06806839
Title: Early Weight Bearing in Distal Femoral Fractures, Dual Plating Versus Single Lateral Plating: a Randomized Controlled Study
Brief Title: Early Weight Bearing in Distal Femur Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Mahmoud Ahmed, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early weight-bearing.
Record Dates: First submitted 2025-01-18; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Distal Femur Fracture
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual plating (Experimental): Participants in this group will undergo dual plating fixation for distal femur fractures.
  Interventions: Procedure: dual plating
- single plating (Active Comparator): Participants in this group will undergo single plate fixation for distal femur fractures.
  Interventions: Procedure: single plating

INTERVENTIONS:
Procedure: dual plating — surgical fixation of the distal femur using two plates to enhance stability and fracture healing.
  Arms: Dual plating
Procedure: single plating — surgical fixation of the distal femur using a single plate according to standard fixation protocols.
  Arms: single plating

SUMMARY:
Assessment of the effect of double plating and single lateral plating on early weight bearing as a primary outcome and improving union and decreasing complications as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients.
* Distal femur fracture type A2, A3, C1, C2 by X-ray (Arbeitsgemeinschaft für Osteosynthesefragen classification).
* Injury Severity Score below 15.
* Controlled comorbidities.
* Fresh fractures: within 3 weeks of trauma.

Exclusion Criteria:

* Distal femur fractures type A1, B, C3 and A2 if there is a medial wedge.
* Open fracture grade 3 Gustilo Anderson Classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Sander's scale. | one year
  A scale of 40 points with 0 as the minimum value and 40 as the maximum value. A higher score means a better outcome. The scale is used as a functional outcome following distal femur fractures fixation using questionaire about the pain, walking ability and return of work and using x rays to measure angulation in degrees and shortening in centimeters and examining the range of motion of the knee joint in degrees.

REFERENCES:
- [Background] Elsoe R, Ceccotti AA, Larsen P. Population-based epidemiology and incidence of distal femur fractures. Int Orthop. 2018 Jan;42(1):191-196. doi: 10.1007/s00264-017-3665-1. Epub 2017 Nov 7. PMID 29116356
- [Background] Myers P, Laboe P, Johnson KJ, Fredericks PD, Crichlow RJ, Maar DC, Weber TG. Patient Mortality in Geriatric Distal Femur Fractures. J Orthop Trauma. 2018 Mar;32(3):111-115. doi: 10.1097/BOT.0000000000001078. PMID 29462121
- [Background] Merino-Rueda LR, Rubio-Saez I, Mills S, Rubio-Suarez JC. Mortality after distal femur fractures in the elderly. Injury. 2021 Jul;52 Suppl 4:S71-S75. doi: 10.1016/j.injury.2021.03.066. Epub 2021 May 5. PMID 33992422
- [Background] Mubark I, Abouelela A, Genena A, Al Ghunimat A, Sarhan I, Ashwood N. Mortality Following Distal Femur Fractures Versus Proximal Femur Fractures in Elderly Population: The Impact of Best Practice Tariff. Cureus. 2020 Sep 30;12(9):e10744. doi: 10.7759/cureus.10744. PMID 33150119
- [Background] Larsen P, Ceccotti AA, Elsoe R. High mortality following distal femur fractures: a cohort study including three hundred and two distal femur fractures. Int Orthop. 2020 Jan;44(1):173-177. doi: 10.1007/s00264-019-04343-9. Epub 2019 May 12. PMID 31081515
- [Background] Poole WEC, Wilson DGG, Guthrie HC, Bellringer SF, Freeman R, Guryel E, Nicol SG. 'Modern' distal femoral locking plates allow safe, early weight-bearing with a high rate of union and low rate of failure: five-year experience from a United Kingdom major trauma centre. Bone Joint J. 2017 Jul;99-B(7):951-957. doi: 10.1302/0301-620X.99B7.BJJ-2016-0585.R1. PMID 28663403
- [Background] Schatzker J, Home G, Waddell J. The Toronto experience with the supracondylar fracture of the femur, 1966-72. Injury. 1974 Nov;6(2):113-28. doi: 10.1016/0020-1383(74)90005-9. No abstract available. PMID 4443073
- [Background] Gangavalli AK, Nwachuku CO. Management of Distal Femur Fractures in Adults: An Overview of Options. Orthop Clin North Am. 2016 Jan;47(1):85-96. doi: 10.1016/j.ocl.2015.08.011. PMID 26614924
- [Background] Atalay IB, Ozturk R, Yapar A, Karakoc Y, Eksioglu MF. Outcomes of the Surgical Treatment of Periprosthetic Fractures Around the Knee with Locking Plates: A Single Centre Experience. Malays Orthop J. 2021 Nov;15(3):1-7. doi: 10.5704/MOJ.2111.001. PMID 34966488
- [Background] Virk JS, Garg SK, Gupta P, Jangira V, Singh J, Rana S. Distal Femur Locking Plate: The Answer to All Distal Femoral Fractures. J Clin Diagn Res. 2016 Oct;10(10):RC01-RC05. doi: 10.7860/JCDR/2016/22071.8759. Epub 2016 Oct 1. PMID 27891409
- [Background] Smith WR, Stoneback JW, Morgan SJ, Stahel PF. Is immediate weight bearing safe for periprosthetic distal femur fractures treated by locked plating? A feasibility study in 52 consecutive patients. Patient Saf Surg. 2016 Dec 7;10:26. doi: 10.1186/s13037-016-0114-9. eCollection 2016. PMID 27980675
- [Background] Striano BM, Grisdela PT Jr, Shapira S, Heng M. Early Weight Bearing after Distal Femur Fracture Fixation. Geriatr Orthop Surg Rehabil. 2022 Jan 27;13:21514593211070128. doi: 10.1177/21514593211070128. eCollection 2022. PMID 35111355
- [Background] Imam MA, Torieh A, Matthana A. Double plating of intra-articular multifragmentary C3-type distal femoral fractures through the anterior approach. Eur J Orthop Surg Traumatol. 2018 Jan;28(1):121-130. doi: 10.1007/s00590-017-2014-9. Epub 2017 Jul 14. PMID 28710534